CLINICAL TRIAL: NCT06049355
Title: EMBark on RAdiation Therapy With a Clinic-based Exercise Program: EXERCISING TOGETHER
Brief Title: EMBRACE: Exercising Together
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Oregon Health and Science University (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Kerri Winters, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY00025294; NCI-2023-02279 (Registry Identifier: CTRP (Clinical Trial Registration Program)); R01CA277738-01 (NIH)
Record Dates: First submitted 2023-09-11; First posted 2023-09-22 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-01

CONDITIONS: Breast Carcinoma; Prostate Carcinoma
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms | interventions — Specimen Handling; Early Intervention, Educational; Educational Status; Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (Exercise Together exercise program) (Experimental): Patients and partners undergo Exercising Together supervised group exercise program using live remote video conference technology over 75 minutes three times a week (TIW) for 8 weeks during radiation therapy on study. Patients also undergo collection of blood samples using self-collection methods throughout the trial.
  Interventions: Other: Exercise Intervention; Procedure: Biospecimen Collection
- Arm II (educational material) (Active Comparator): Patients and partners receive educational materials specific to exercise. Patients also undergo collection of blood samples using self collection methods throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Other: Educational Intervention

INTERVENTIONS:
Other: Exercise Intervention — Undergo Exercise Together exercise program, a supervised group exercise program delivered online, using a live remote format
  Arms: Arm I (Exercise Together exercise program)
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection, Biological Sample Collection, Biospecimen Collected, Biospecimen Collection, Specimen Collection
Other: Educational Intervention — Receive educational materials
  Other Names: Education for Intervention, Intervention by Education, Intervention through Education, Intervention, Educational
  Arms: Arm II (educational material)

SUMMARY:
This phase II trial tests how well an exercise intervention, Exercising Together, works in preventing declines in physical and mental health in couples during radiation treatment for cancer. Treatments for cancer can cause side effects such as fatigue as well as strain on relationships. Exercising Together is a partnered exercise program that adds communication, collaboration and support between partners during exercise to fortify the relationship and amplify the benefits of physical training. Exercising Together program may be effective on the mental and physical health of couples during radiation treatment for cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To test the effectiveness and mechanisms of the adapted Exercise Together intervention on mental and physical health of couples (Aims 1 & 2).

SECONDARY OBJECTIVE:

I. To gain better understanding of the implementation context and implementation outcomes (Aim 3).

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients and partners undergo Exercising Together exercise program during radiation therapy on study. Patients also undergo collection of blood samples throughout the trial.

ARM II: Patients and partners receive educational materials specific to exercise. Patients also undergo collection of blood samples throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

* INTERVENTION (SURVIVORS) INCLUSION

  * Histologically confirmed prostate cancer or breast cancer without evidence of metastatic disease
  * Confirmed by review of the electronic medical record (EMR) and subsequently recorded in Survivor Health History. In cases where the EMR isn't clear, their Oregon Health & Science University (OHSU) provider will be contacted for confirmation. For non-OHSU patients, we'll initially collect their cancer health history by a self-report questionnaire and confirm when we receive the survivor's outside medical record (through a signed Release of Information)
* Scheduled to receive radiation therapy for curative intent

  * Confirmed by review of the EMR and subsequently recorded in Survivor Health History. In cases where the EMR isn't clear, their OHSU provider will be contacted for confirmation/ For non-OHSU patients, we'll initially collect their cancer health history by a self-report questionnaire and confirm when we receive the survivor's outside medical record (through a signed Release of Information)
* Co-residing with an intimate partner or spouse who is willing to participate

  * Confirmed by self-report on the Demographic Questionnaire
* INTERVENTION (SURVIVORS AND PARTNERS) INCLUSION
* 18 years of age and older

  * For survivors: confirmed by review of the date of birth as documented in the Electronic Medical Record (EMR) and subsequently recorded in Survivor Health History. For non-OHSU patients, we'll collect their age by self-report on the Survivor Health History
  * For partners: confirmed by self-report on the Health History Questionnaire
* < 2 structured strength training sessions for less than 30 minutes per week in the last month

  * Confirmed by self-report on Health History Questionnaire
* Home internet sufficient for videoconferencing

  * Confirmed by staff review of Internet Connectivity Screening Guide with the participants and outcome recorded in a CRF
* Signed informed consent

  * Confirmed by completion of e-Consent in REDCap
* Willing to be randomized into either study arm and adhere to study protocol

  * Confirmed verbally with the participant and response documented in the Participant Tracking database
* IMPLEMENTATION INCLUSION
* Be one of these key stakeholders: patient, spouse/partner, healthcare providers, or administrator
* Verbal informed consent following receipt of an Information Sheet

Exclusion Criteria:

* INTERVENTION (SURVIVORS AND PARTNERS) EXCLUSION
* Cognitive difficulties that preclude answering the survey questions, participating in the exercise classes or performance tests, or providing informed consent

  * In the event of a suspected undeclared cognitive impairment, it will be confirmed by physician clearance or professional opinion of the Principal Investigator, Kerri Winters-Stone
* A medical condition, movement or neurological disorder, or medication use that contraindicates participation in moderate intensity exercise. Specific contraindications include the following: poorly controlled diabetes, recent cardiac event, neuromuscular disease, untreated orthostatic hypertension, recent surgery, acute hernia, acute rheumatoid arthritis, severe memory disorders, severe balance disorder, inability to ambulate without a walker or wheelchair, inability to stand for 3 minutes, severe hearing or vision problem

  * Confirmed by a combination of reviewing the EMR, self-report on the Health History Questionnaire, Charlson Comorbidity Index questionnaire, and/or by physician clearance. If in the professional opinion of the Principal Investigator, Dr. Kerri Winters-Stone, contraindications other than those identified by the patient or physician are present, she may consider the participant ineligible. For Spouse/Partner: must answer 'No' to American College of Sports Medicine pre-participation screening questions. If spouse/partner answers 'Yes' to either question they may be required to obtain physician clearance prior to becoming eligible. Physician clearance may also be requested at the discretion of the principal investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-04-18 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Physical functioning | Baseline, Months 2, Month 4, and Month 6
  Measured by the Physical Performance Battery (PPB) to determine a person's ability to perform daily tasks independently. The PPB consists of 3 timed tests: 5 repeated chair stands, standing balance, and usual pace gait speed over 4 meters. Each test is scored 0 (unable) to 4 (completes without difficulty), based on quartiles of performance, then scores are summed. The possible range of scores is 0-12.
Anxiety | Baseline, Month 1, Month 2, Month 4, and Month 6
  Measured by the Patient Reported Outcomes Measurement Information System (PROMIS) anxiety short form using questions on a scale ranging from 1 (never) to 5 (always).

SECONDARY OUTCOMES:
Changes in patient-reported symptoms | Baseline, Month 1, Month 2, Month 4, and Month 6
  Measured by PROMIS to assess symptoms of physical and mental health and global health (QoL). We will use the 13-item measure and 8-item measures for symptoms in the past 7 days. Global health is assessed with a 10-item measure that asks about physical, mental and social functioning.
Sexual function and satisfaction | Baseline, Month 1, Month 2, Month 4, and Month 6
  Assessed with a 14-item measure in the past 30 days and is specific to either male or female
Sleep Behavior: total sleep time | Baseline, Months 2, Month 4, and Month 6
  Measured using ActiGraph Link, we will have extended wear time to measures total sleep time over a 3-day monitoring period.
Inflammation - high sensitivity C-Reactive Protein (hsCRP) | Baseline, Months 2, and Month 6
  Measured using a self-administered dried blood spot (DBS) collection kit. Participants are taught by research staff and follow a YouTube video to use a finger stick poke to obtain a drop of blood that is put onto a sample card. DBS captured on the designated card are dried thoroughly (> 4 hours at room temperature), then inserted into a foil pouch with desiccant and mailed to the research team. Cards are frozen (0 degree Fahrenheit [F] or below) until analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Kerri Winters-Stone, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual quantitative participant data collected during the trial, after deidentification.
Time Frame: Beginning 3 months following final publication.
Access Criteria: Access will be provided to investigators who provide a methodologically sound proposal and complete a data sharing agreement that includes commitments to: (1) using the data only for research purposes and not to identify any individual participant, (2) securing the data using appropriate computer technology, and (3) destroying or returning the data after analyses are completed.
  Proposals should be directed to wintersk@ohsu.edu. To gain access to data, data requestors will need to sign a data sharing agreement.